CLINICAL TRIAL: NCT04693546
Title: Subject Enrollment and Specimen Collection Protocol to Validate the Performance of the LifeKit® Prevent Colorectal Neoplasia Test for Colorectal Cancer Screening
Brief Title: Protocol to Validate the Performance of the LifeKit® Prevent Colorectal Neoplasia Test for CRC Screening
Acronym: PREVENT
Status: Suspended | Type: Observational
Why Stopped: fundraising
Sponsor: Metabiomics Corp (Industry)
Responsible Party: Sponsor
Other Study IDs: PM-2020-001
Record Dates: First submitted 2020-12-28; First posted 2021-01-05 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer; Colorectal Adenoma
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: LifeKit Prevent Colorectal Neoplasia Test — Procedure: Colonoscopy
Diagnostic Test: FIT Test — Procedure: Colonoscopy

SUMMARY:
The purpose of this study is to determine the sensitivity and specificity for LifeKit Prevent Colorectal Neoplasia Test for colorectal cancer (CRC) and for adenoma, including advanced adenoma.

DETAILED DESCRIPTION:
Subjects 40 years of age and older scheduled for a screening colonoscopy will be enrolled. Subjects will collect a stool sample that will be tested by the LifeKit Prevent Colorectal Neoplasia Test at a central laboratory and that will be tested using a commercially available FIT. After sample collection, subjects will undergo a screening colonoscopy per standard of care. Investigators will be blinded to the results of the LifeKit Prevent Colorectal Neoplasia Test during the study; the LifeKit Prevent Colorectal Neoplasia Test and FIT results will not be used for clinical management of subjects. Personnel performing the colonoscopy and reports from the colonoscopy and personnel performing the histopathological review of the tissue and/or any reports will remain blinded to the results of the LifeKit Prevent Colorectal Neoplasia Test results.

ELIGIBILITY:
Inclusion Criteria:

An individual must meet all of the criteria below to be eligible.

1. Subject is ≥ 40 years of age at the time of enrollment.
2. Subject presents for a screening colonoscopy per standard of care.
3. Subject has no symptoms or signs that require immediate, or near term, referral for diagnostic or therapeutic colonoscopy.
4. Subject is able and willing to sign informed consent.

Exclusion Criteria:

An individual meeting any of the below criteria is ineligible.

1. Subject has a history of CRC or advanced precancerous lesions.
2. Subject has a diagnosis or medical history of any of the following conditions:

   * Familial adenomatous polyposis (also referred to as "FAP", including attenuated FAP and Gardner's syndrome)
   * Hereditary non-polyposis CRC syndrome (also referred to as "HNPCC" or "Lynch Syndrome")
   * Other hereditary cancer syndromes, including but are not limited to, Peutz-Jeghers Syndrome, MYH-Associated Polyposis (MAP), Turcot's (or Crail's) Syndrome, Cowden's Syndrome, Juvenile Polyposis, Neurofibromatosis, or Familial Hyperplastic Polyposis
3. Subject has a diagnosis or personal history of inflammatory bowel disease (IBD), including chronic ulcerative colitis or Crohn's disease.
4. Subject has a diagnosis of Cronkhite-Canada Syndrome.
5. Subject has had a positive Cologuard, fecal occult blood test or FIT within the previous 2 years.
6. Subject has undergone a colonoscopy within the previous 9 years.
7. Subject has had overt rectal bleeding within the previous 30 days.
8. Subject has any condition that in the opinion of the Investigator should preclude participation in the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects 40 years of age and older who are eligible for colorectal cancer screening and scheduled for a screening colonoscopy per standard of care. Approximately 12,000 subjects will be targeted for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity for the LifeKit Prevent Colorectal Neoplasia Test for adenoma, including advanced adenoma | Through study completion, an average of 180 days

SECONDARY OUTCOMES:
Sensitivity and specificity of the LifeKit Prevent Colorectal Neoplasia Test for colorectal cancer | Through study completion, an average of 180 days
Sensitivity and specificity of the LifeKit Prevent Colorectal Neoplasia Test for advanced adenoma | Through study completion, an average of 180 days
Sensitivity of the LifeKit Prevent Colorectal Neoplasia Test is non-inferior to that of FIT for colorectal cancer | Through study completion, an average of 180 days
Sensitivity of the LifeKit Prevent Colorectal Neoplasia Test is superior to that of FIT for advanced adenoma | Through study completion, an average of 180 days

CONTACTS AND LOCATIONS:
Locations (1):
- Solvd Health, Carlsbad, California, United States